CLINICAL TRIAL: NCT00640432
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Study Of The Safety, Tolerability And Efficacy Of Celecoxib 200 Mg Twice A Day (With A 400 Mg Attack Dose) Versus Sodium Diclofenac 75 Mg Twice A Day In Subjects With Acute Low Back Pain
Brief Title: Safety And Efficacy Of Celecoxib Versus Sodium Diclofenac In The Treatment Of Acute Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191064
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Diclofenac; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Diclofenac
- B (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Diclofenac — 75 mg oral capsule twice daily for 7 days
  Arms: A
Drug: Celecoxib — 400 mg oral capsule followed by 200 mg oral capsule with the evening meal (>=4 hours from first dose) on Day 1 then 200 mg oral capsule twice daily for 6 days
  Arms: B

SUMMARY:
To evaluate the safety and efficacy of celecoxib versus sodium diclofenac in subjects with acute low back pain

ELIGIBILITY:
Inclusion criteria:

* Aged between 18 and 65 years
* Acute low back pain that falls into 1st or 2nd class of 'Quebec Task Force' classification of moderate to severe intensity (>50 mm in the VAS)
* Acute low back pain onset <72 hours prior to study inclusion and >6 weeks after the last acute low back pain episode

Exclusion criteria:

* Scoliosis or known history of inflammatory arthritis, chronic pain, metastasis, Paget's disease, or any other disease that cause pain
* Low back pain from major trauma or visceral disorder
* Esophageal ulcers, gastric or duodenal ulcers or bleeding within 30 days prior to being administered study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2003-10; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient-rated visual analogue scale (VAS) pain intensity assessment | Day 3

SECONDARY OUTCOMES:
Subject's quality of life, as measured by the SF-36 Health Survey | Day 7
Physical examination | Days 3 and 7
Pain relief score | Days 3 and 7
Vital signs | Days 3 and 7
Adverse events | Days 3 and 7
Change from baseline in VAS pain intensity assessment | Day 7
Categorical pain intensity score | Days 3 and 7
Subject's global assessment score | Days 3 and 7
Subject's functional ability, as measured by the "Roland Morris" Questionnaire about low back pain and disability | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Brazil (5):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Londrina, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191064&StudyName=Safety%20And%20Efficacy%20Of%20Celecoxib%20Versus%20Sodium%20Diclofenac%20In%20The%20Treatment%20Of%20Acute%20Low%20Back%20Pain